CLINICAL TRIAL: NCT04174144
Title: The Effect of Lordosis on Long-term Clinical Outcome and Sagittal Balance Parameters After TLIF for One-level Degenerative Spondylolysthesis
Brief Title: The Effect of Lordosis on Clinical Outcome After Spinal Fusion for One-level Degenerative Spondylolysthesis
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Klemen Bošnjak, Resident of Orthopaedic surgery, University Medical Centre Ljubljana
Other Study IDs: 0120-259/2019/6
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Spondylolisthesis Degenerative; Spinal Fusion
Keywords: Sagittal balance; Lumbar lordosis; Clinical outcomes
MeSH Terms: conditions — Lordosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TLIF group: Participants with degenerative spondylolysthesis who underwent a single-level TLIF procedure.
  Interventions: Procedure: Single-level TLIF

INTERVENTIONS:
Procedure: Single-level TLIF — Transforaminal interbody fusion approach, using polyaxial pedicle screws (Xia®, Stryker Spine, Allendale, NJ, USA), combined with a crescent-shaped interbody cage (T-Plus®, Pioneer Surgical Technology, Marquette, MI, USA), bilateral facet joint removal and laminectomy.

SUMMARY:
Degenerative spondylolisthesis is a common spinal degenerative disease. It is defined as the slippage of one vertebrae on the vertebrae bellow. In the process of spinal ageing and spinal joint degeneration, the spine becomes subjected to degenerative development that results in joint instability, shifting of vertebrae and can be responsible for a progressive kyphosis of the lumbar spine and sagittal imbalance with forward inclination of the trunk and chronic low back pain development. To address these changes and restore stability, lumbar spinal fusion has been developed and is nowadays a common procedure for unstable degenerative spine disorders.

In the past several years, studies that highlight the importance of sagittal balance analysis with the restoration of adequate lumbar lordosis, have emerged. However, it remains a challenge to determine the correct amount of lumbar lordosis that is required for each patient to maintain optimal post-fusion sagittal balance. Additionally, the relationship between pelvic incidence (PI) and impact of LL correction has been highlighted in literature. The position of fused vertebrae is of paramount importance, as sagittal alignment should be done with minimizing muscle work during posture. Failure to reach proper sagittal balance can result in compensatory mechanisms such as increased pelvic tilt (PT), cervical and thoracic segment hyperextension, and knee flexion. These compensatory mechanisms have adverse effects such as chronic pain, disability and muscle fatigue.

With this study the investigators aim to analyze long-term clinical and spinopelvic radiographic parameter outcomes of patients who underwent a one-level spinal fusion procedure for single level degenerative spondylolisthesis disease at a single institution.

DETAILED DESCRIPTION:
TLIF (transforaminal interbody fusion) is a safe and effective treatment option for single-level lumbar degenerative disease. It is less invasive, yields good outcomes and has fewer complications after long-term follow up compared to other fusion techniques. In literature, many studies have compared sagittal parameters and functional outcomes in single-level TLIF surgery. In most literature reports, however, the fusion was performed at different lumbar levels, depending on the characteristics of the studied cohort. As demonstrated by Roussouly et. al. in the asymptomatic population, the L4 vertebra represents the apex of lumbar lordosis and is the most suitable site for lordosis correction. There are several reported surgical techniques and methods to obtain adequate lordosis correction during TLIF.

At Department of Orthopaedic surgery of Ljubljana University medical centre, TLIF is performed using a consistent brand of instrumentation. In knee-chest position, polyaxial pedicle screws (Xia®, Stryker Spine, Allendale, NJ, USA), combined with a crescent-shaped interbody cage (T-Plus®, Pioneer Surgical Technology, Marquette, MI, USA), bilateral facet joint removal and laminectomy on both sides are used. Compression over the rods is performed to obtain adequate segmental lordosis. The angle of lordosis correction is calculated according Schwab's formula (ideal lumbar lordosis (LL) = pelvic incidence (PI) + 9).

There is little published information regarding cohorts with long-term evaluation. As many authors suggested, changes in lordotic parameters can become clinically evident several years after the procedure. With this study's cohort analysis, a rarely reported link between spinopelvic parameters and long-term clinical evaluation will be demonstrated. Selected participants will be analyzed using the same protocol as preoperatively. A clinical examination will be made, ODI questionnaires will be administered and radiographic parameters on full-standing lateral radiographs, will be analyzed. Changes between preoperative and long-term postoperative parameters will be calculated and compared. For statistical analysis paired t-test and Pearson correlation will be used. All statistical tests will be two tailed and significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one-level degenerative spondylolysthesis treated with single-level TLIF at Department of Orthopaedic surgery of Ljubljana University medical centre between 2011 and 2013.
* TLIF performed at L3/4 or L4/5

Exclusion Criteria:

* Patients who refuse to participate in study or do not respond to our invitation
* Patients with additional instrumental spinal surgery or spinal trauma
* Patients with additional types of adult spinal deformity
* Patients with inflammatory spinal conditions
* Patients with flexion contractures of the hips or knees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients who underwent a single-level TLIF procedure at Department of Orthopaedic surgery of Ljubljana University medical centre between 2011 and 2013.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
ODI questionnaire | 7-9 years after TLIF procedure
  The Oswestry Disability Index is an important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. For each section the total possible score is 5. If all 10 sections are completed the maximal score is 50.
LL | 7-9 years after TLIF procedure
  Radiographic evaluation of lumbar lordosis (LL): the angle between the upper endplate of the first lumbar vertebrae (L1) and the sacral endplate (S1).
SL | 7-9 years after TLIF procedure
  Radiographic evaluation of segmental lordosis (SL): the angle between the cranial endplate of the upper and caudal endplate of the lower vertebrae of the operated segment.

SECONDARY OUTCOMES:
PT | 7-9 years after TLIF procedure
  Radiographic evaluation of pelvic tilt (PT): the angle between the vertical line and the line going through the middle of the femoral heads and the middle point of the sacral endplate.
SS | 7-9 years after TLIF procedure
  Radiographic evaluation of sacral slope (SS): the angle between sacral endplate and the horizontal line.
SVA | 7-9 years after TLIF procedure
  Radiographic evaluation of sagittal vertical axis (SVA): a horizontal distance between the posterior end of the sacral endplate and the vertical line extended through the middle of seventh cervical vertebrae.

CONTACTS AND LOCATIONS:
Overall Officials: Rok Vengust, M.D, PhD, Study Chair — Department of Orthopaedic surgery, University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication and are in accordance with ethical standards of the National ethics committee of Slovenia on human experimentation and with the Helsinki Declaration of 1975.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting within 1 year after publication.
Access Criteria: IPD and any additional supporting information will be shared by request with the Principal investigator.

REFERENCES:
- [Background] Barrey C, Roussouly P, Le Huec JC, D'Acunzi G, Perrin G. Compensatory mechanisms contributing to keep the sagittal balance of the spine. Eur Spine J. 2013 Nov;22 Suppl 6(Suppl 6):S834-41. doi: 10.1007/s00586-013-3030-z. Epub 2013 Sep 20. PMID 24052406
- [Background] Barrey C, Darnis A. Current strategies for the restoration of adequate lordosis during lumbar fusion. World J Orthop. 2015 Jan 18;6(1):117-26. doi: 10.5312/wjo.v6.i1.117. eCollection 2015 Jan 18. PMID 25621216
- [Background] Cheng X, Zhang F, Zhang K, Sun X, Zhao C, Li H, Li YM, Zhao J. Effect of Single-Level Transforaminal Lumbar Interbody Fusion on Segmental and Overall Lumbar Lordosis in Patients with Lumbar Degenerative Disease. World Neurosurg. 2018 Jan;109:e244-e251. doi: 10.1016/j.wneu.2017.09.154. Epub 2017 Oct 5. PMID 28987851
- [Background] Ferrero E, Ould-Slimane M, Gille O, Guigui P; French Spine Society (SFCR). Sagittal spinopelvic alignment in 654 degenerative spondylolisthesis. Eur Spine J. 2015 Jun;24(6):1219-27. doi: 10.1007/s00586-015-3778-4. Epub 2015 Feb 5. PMID 25652553
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Kuhta M, Bosnjak K, Vengust R. Failure to maintain segmental lordosis during TLIF for one-level degenerative spondylolisthesis negatively affects clinical outcome 5 years postoperatively: a prospective cohort of 57 patients. Eur Spine J. 2019 Apr;28(4):745-750. doi: 10.1007/s00586-019-05890-w. Epub 2019 Jan 24. PMID 30680634
- [Background] Le Huec JC, Aunoble S, Philippe L, Nicolas P. Pelvic parameters: origin and significance. Eur Spine J. 2011 Sep;20 Suppl 5(Suppl 5):564-71. doi: 10.1007/s00586-011-1940-1. Epub 2011 Aug 10. PMID 21830079
- [Background] Le Huec JC, Faundez A, Dominguez D, Hoffmeyer P, Aunoble S. Evidence showing the relationship between sagittal balance and clinical outcomes in surgical treatment of degenerative spinal diseases: a literature review. Int Orthop. 2015 Jan;39(1):87-95. doi: 10.1007/s00264-014-2516-6. Epub 2014 Sep 6. PMID 25192690
- [Background] Le Huec JC, Hasegawa K. Normative values for the spine shape parameters using 3D standing analysis from a database of 268 asymptomatic Caucasian and Japanese subjects. Eur Spine J. 2016 Nov;25(11):3630-3637. doi: 10.1007/s00586-016-4485-5. Epub 2016 Mar 7. PMID 26951168
- [Background] Liang Y, Shi W, Jiang C, Chen Z, Liu F, Feng Z, Jiang X. Clinical outcomes and sagittal alignment of single-level unilateral instrumented transforaminal lumbar interbody fusion with a 4 to 5-year follow-up. Eur Spine J. 2015 Nov;24(11):2560-6. doi: 10.1007/s00586-015-3933-y. Epub 2015 Apr 14. PMID 25870077
- [Background] Morvan G, Mathieu P, Vuillemin V, Guerini H, Bossard P, Zeitoun F, Wybier M. Standardized way for imaging of the sagittal spinal balance. Eur Spine J. 2011 Sep;20 Suppl 5(Suppl 5):602-8. doi: 10.1007/s00586-011-1927-y. Epub 2011 Aug 10. PMID 21830081
- [Background] Ould-Slimane M, Lenoir T, Dauzac C, Rillardon L, Hoffmann E, Guigui P, Ilharreborde B. Influence of transforaminal lumbar interbody fusion procedures on spinal and pelvic parameters of sagittal balance. Eur Spine J. 2012 Jun;21(6):1200-6. doi: 10.1007/s00586-011-2124-8. Epub 2011 Dec 17. PMID 22179755
- [Background] Roussouly P, Pinheiro-Franco JL. Biomechanical analysis of the spino-pelvic organization and adaptation in pathology. Eur Spine J. 2011 Sep;20 Suppl 5(Suppl 5):609-18. doi: 10.1007/s00586-011-1928-x. Epub 2011 Aug 2. PMID 21809016
- [Background] Schwab F, Lafage V, Patel A, Farcy JP. Sagittal plane considerations and the pelvis in the adult patient. Spine (Phila Pa 1976). 2009 Aug 1;34(17):1828-33. doi: 10.1097/BRS.0b013e3181a13c08. PMID 19644334
- [Background] Tye EY, Alentado VJ, Mroz TE, Orr RD, Steinmetz MP. Comparison of Clinical and Radiographic Outcomes in Patients Receiving Single-Level Transforaminal Lumbar Interbody Fusion With Removal of Unilateral or Bilateral Facet Joints. Spine (Phila Pa 1976). 2016 Sep;41(17):E1039-E1045. doi: 10.1097/BRS.0000000000001535. PMID 26926356